CLINICAL TRIAL: NCT01799408
Title: The Effect of Intra-articular Injection of Betamethasone Acetate/Betamethasone Sodium Phosphate at the Knee Joint on the Hypothalamic-pituitary-adrenal Axis: a Case Controlled Study
Brief Title: Intra-articular Betamethasone and the Hypothalamic-pituitary-adrenal Axis
Status: Completed | Type: Observational
Sponsor: The Nazareth Hospital, Israel (Other)
Responsible Party: Principal Investigator, George Habib, Head rheunatology clinic, The Nazareth Hospital, Israel
Other Study IDs: HPA-2012
Record Dates: First submitted 2013-02-21; First posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Adrenal Suppression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- betamethasone: Patients who had intra-articular injection of betamethasone
- Hyaluronic acid: Patients who had intra-articular injection of hyaluronic acid

SUMMARY:
To evaluate the effect of intra-articular corticosteroid injection (IACI) of depot preparation of betamethasone on the hypothalamic-pituitary-adrenal (HPA) axis, in patients with osteoarthritis of the knee

DETAILED DESCRIPTION:
Consecutive patients attending the rheumatology or orthopedic clinic with osteoarthritic knee pain, not responding satisfactorily to medical or physical therapy were allocated to group-1 after consent and given IACI of 6 mg of betamethasone acetate/betamethasone sodium phosphate. Following completion of this part, consecutive age- and sex-matched patients were allocated to group-2 and given intra-articular injection of 60 mg of sodium hyaluronate. Just prior to the knee injection and 1, 2, 3, 4 and 8 weeks later, patients had 1 µg adrenocorticotropin hormone (ACTH) stimulation test. Secondary adrenal insufficiency (SAI) was defined as levels of less than 18 ng/ml or a rise of < than 7 ng/ml of serum cortisol, 30 minutes following the ACTH stimulation test.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee

Exclusion Criteria:

* Had steroids in the last 3 months. Allergic to steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with osteoarthritis of the knee and had not been onsteroids for at least 3 months
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Adrenal Suppression | 2 months
  Adrenal gland suupresion and inability to adequately secrete cortisol in response to stress

SECONDARY OUTCOMES:
favorable clinical response | 2 months
Favorable clinical response | 2 months following the steroid injection
  Improvement of knee pain by more than 30 points according to visual analogue scale

OTHER OUTCOMES:
Nadir serum cortisol level | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: George Habib, M.D., Principal Investigator — Nazareth Hospital